CLINICAL TRIAL: NCT05486962
Title: Remote Monitoring of Surgical Patients Through VALIDIC
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00110616
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Elective Abdominal Surgery
MeSH Terms: interventions — Remote Patient Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Remote Patient Monitoring: Patients undergoing elective abdominal surgery will be asked to use a wearable activity tracker, vivosmart®HR by Garmin, pre and post-operatively to help remotely monitor health metrics. Data collected through the Garmin device will be reviewed to assess compliance and improvement in activity. Aggregate data will be analyzed to assess feasibility and effectiveness of this device in improving patient recovery.
  Interventions: Behavioral: Remote Patient Monitoring

INTERVENTIONS:
Behavioral: Remote Patient Monitoring — Patients undergoing elective abdominal surgery will be asked to use a wearable activity tracker, vivosmart®HR by Garmin, pre and post-operatively to help remotely monitor health metrics. Data collected through the Garmin device will be reviewed to assess compliance and improvement in activity. Aggregate data will be analyzed to assess feasibility and effectiveness of this device in improving patient recovery.
  Other Names: vivosmart®HR; VALIDIC

SUMMARY:
We propose to assess the feasibility and outcomes of use of a wearable activity tracker for monitoring daily step counts in the peri-operative and 30 day post-operative period in elderly patients receiving elective abdominal surgery at Duke. We will use the information as guidance for improving activity in surgical patients at Duke. The activity tracker will be worn for the peri-operative period which starts at the time of the surgery/clinic visit and continues during the inpatient hospital stay and for 30 days following discharge. The vivosmart®HR is a commercially available device that is made of plastic and designed to be worn around the wrist. Aggregate data will be analyzed to assess feasibility and effectiveness of this device in improving patient recovery. No discomfort or burden is expected from wearing the monitor, and patients will have continuous feedback on their daily activity.

DETAILED DESCRIPTION:
We propose to assess the feasibility and outcomes of use of a wearable activity tracker for monitoring daily step counts in the peri-operative and 30 day post-operative period in elderly patients receiving elective abdominal surgery at Duke. We will use the information as guidance for improving activity in surgical patients at Duke. All ambulatory patients going through the POSH program currently receive individualized counseling on enhancing their activity levels. The data collected in this project will be used to help refine counseling and identify optimal time frames where exercise counseling is most beneficial. Our goal is to help with disease management, remote monitoring alerts, readmission prevention, care coordination and placement of required consults.

Aim1: Evaluate the feasibility of data capture, data integration into EPIC, and validate data flow Aim 2: Retrospective review of data to identify opportunities for alerts Aim 3: Improve physical function of older patients

This is a prospective remote patient monitoring study in the peri-operative and post-operative period to improve surgical outcomes. The peri-operative period starts at the time of the surgery/POSH clinic visit, continues during the inpatient hospital stay and for 30 days following discharge.

Patients undergoing elective abdominal surgery will be asked to use a wearable activity tracker, vivosmart®HR by Garmin, pre and post-operatively to help remotely monitor health metrics. Data collected through the Garmin device will be reviewed to assess compliance and improvement in activity. Aggregate data will be analyzed to assess feasibility and effectiveness of this device in improving patient recovery. The metrics we plan to assess are the following:

Garmin data:

Steps, distance, calories, heart rate, 7 day resting average, floors climbed activity intensity, sleep cycles, inactive periods.

Surgery data:

Length of stay, Complications, Readmissions, Emergency Department visits

Patients may be called weekly to ensure compliance and ask any questions or report any issues with the activity tracker. All data will exist in MaestroCare and will be captured after the post-surgical period.

ELIGIBILITY:
Inclusion Criteria:

1. Over 75 yo
2. HBP procedures, Colorectal procedures, Open VHRs
3. No obvious cognitive deficits
4. Should be able to walk with or without mobility aid
5. Willingness to use smart phone in the study

Exclusion Criteria:

1. non-ambulatory status,
2. dementia, or
3. a pending cardiac clearance requirement for surgery.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients undergoing elective abdominal surgery at Duke.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Enrollment
  proportion of those who were approached and eligible, and who agreed to participate (i.e., recruitment rates)
Completion Rate | 30 days post-operatively
  proportion of those who completed the protocol (i.e., completion rate)
Retention Rate | 30 days post-operatively
  proportion who participated in all three settings (pre hospital, hospital, post hospital) (i.e., retention rate),
Scale-Level Completion Rate | 30 days post-operatively
  proportion who completed use of the activity trackers, and determine the reason for any missing data including lack of understanding, ability, or simple refusal (i.e., scale-level completion rate);
Study Duration | 45 days after last patient enrollment
  documented duration of the protocol (i.e., feasibility);

SECONDARY OUTCOMES:
Alert Timepoints | 30 days post-operatively
  Retrospective review of data to identify opportunities for alerts:
  LOS, Complications, Readmissions, ED visits
Physical Function | 30 days post-operatively
  Improve physical function of older patients by evaluating:
  LOS, Complications, Readmissions, ED visits

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya Lagoo-Deenadayalan, MD, PhD, Principal Investigator — Duke Medical Center
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No